CLINICAL TRIAL: NCT06863454
Title: Trichoscopy as a Monitoring Tool for Activity and Remission in Pemphigus Vulgaris: A Clinical Study Supported by Immunological Evaluation.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Abd El-nasser Attay, Principle investigator, Assiut University
Other Study IDs: Tricho PV
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Pemphigus Vulgaris (PV)
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: cases of PV with disease activity
  Interventions: Diagnostic Test: Trichoscopy
- Group 2: cases of PV with disease remission
  Interventions: Diagnostic Test: Trichoscopy
- Group 3: control group

INTERVENTIONS:
Diagnostic Test: Trichoscopy — Trichoscopy will be done on patients with PV disease activity and remission
  Groups: Group 1; Group 2

SUMMARY:
Pemphigus vulgaris (PV) is a potential life-threatening autoimmune bullous disorder presenting with multiple erosions and flaccid blisters that can involve both mucous membrane and skin. The microscopic findings include intraepithelial blisters caused by acantholysis of keratinocytes as the consequence of autoantibody formation. The antibodies are mainly IgG autoantibodies mostly directed against desmoglein 1 and 3 (Dsg 1, 3), which are adhesion molecules expressed on the surface of keratinocytes.

DETAILED DESCRIPTION:
Scalp is a unique location for pemphigus because of the abundance of desmogleins localized in hair follicles. The frequency of scalp involvement in the course of pemphigus is estimated at 16-60% . According to literature data, the scalp is the first location in 9-15% of patients with pemphigus.

Several cases of alopecia in the course of pemphigus have been described. The significance of the distribution of desmogleins in hair follicles for scalp involvement and a potential use of direct immunofluorescence of plucked hairs are discussed in the literature. The significance of scalp involvement for the course of pemphigus remains controversial.

Trichoscopy is a non-invasive method for diagnosing hair and scalp disorders. Trichoscopy is widely used to differentiate causes of scalp lesions and scarring and non-scarring alopecia. To date there are few studies on the value of trichoscopy in pemphigus.

The pathogenesis and pathophysiology of PV depend on various factors like cellular immunity, genetic factors, ethnicity, diet and environment. According to previous studies, Dsg autoantibodies with IgG1 and IgG4 subtypes are mostly detected in the active form of the pemphigus diseases. Accordingly, the significant role of autoreactive B cells in the pathogenesis of PV could be explained by producing these types of autoantibodies.

Recently attention has been directed toward the role of T cells in the pathogenesis of PV. Similar to other autoimmune diseases, the underlying etiology of PV depends on the interaction between T cells and B cells resulting in antibody secretion.

Autoreactive CD4+ T cells are essential for the pathogenesis of several ab-mediated autoimmune diseases by providing help to autoreactive B cells resulting in the production of antigen specific auto-ab. Alterations in several T cell subsets like CD4+CD25+ Treg and Th17 cells, have been described and are suggested to play a role in the pathogenesis of pemphigus.

A few studies have investigated the significant role of T cell subgroups, namely regulatory T cells (Treg), T helper17 (Th17), and T follicular helper cells (Tfh) in PV and some studies were carried out on both human and mouse models to meticulously reveal the function of T cell phenotypes including CD8+T cells, γδ T cells, and resident memory T cells in the pathogenesis of PV, which may explain the wide range of clinical presentations and severity of PV in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and histopathological diagnosis of pemphigus vulgaris will be included.
* Pemphigus patients are categorized as active or remittent.

Exclusion Criteria:

* Other forms of pemphigus.
* Patients who are previously treated with rituximab.
* Patients with any concomitant dermatological diseases.
* Patients with other autoimmune diseases.
* Pregnancy and lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from those attending the Bullous outpatient clinic of department of Dermatology, Assiut University Hospitals with the diagnosis of pemphigus vulgaris. Patients will be included in the study after obtaining a written informed consent. And after the approval of the faculty of medicine ethics committee. An age and sex matched healthy volunteers will be recruited as a control group.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Trichoscopy as a monitooring tool | 1 year
  for activity and remission in PV

REFERENCES:
- [Background] Xu RC, Zhu HQ, Li WP, Zhao XQ, Yuan HJ, Zheng J, Pan M. The imbalance of Th17 and regulatory T cells in pemphigus patients. Eur J Dermatol. 2013 Nov-Dec;23(6):795-802. doi: 10.1684/ejd.2013.2177. PMID 24192290
- [Background] Wu H, Stanley JR, Cotsarelis G. Desmoglein isotype expression in the hair follicle and its cysts correlates with type of keratinization and degree of differentiation. J Invest Dermatol. 2003 Jun;120(6):1052-7. doi: 10.1046/j.1523-1747.2003.12234.x. PMID 12787134
- [Background] Veraitch O, Ohyama M, Yamagami J, Amagai M. Alopecia as a rare but distinct manifestation of pemphigus vulgaris. J Eur Acad Dermatol Venereol. 2013 Jan;27(1):86-91. doi: 10.1111/j.1468-3083.2011.04363.x. Epub 2011 Nov 28. PMID 22122058
- [Background] Tavakolpour S, Mahmoudi H, Mirzazadeh A, Balighi K, Darabi-Monadi S, Hatami S, GhasemiAdl M, Daneshpazhooh M. Pathogenic and protective roles of cytokines in pemphigus: A systematic review. Cytokine. 2020 May;129:155026. doi: 10.1016/j.cyto.2020.155026. Epub 2020 Feb 10. PMID 32058276
- [Background] Takahashi H, Amagai M, Nishikawa T, Fujii Y, Kawakami Y, Kuwana M. Novel system evaluating in vivo pathogenicity of desmoglein 3-reactive T cell clones using murine pemphigus vulgaris. J Immunol. 2008 Jul 15;181(2):1526-35. doi: 10.4049/jimmunol.181.2.1526. PMID 18606708
- [Background] Sar-Pomian M, Rudnicka L, Olszewska M. The Significance of Scalp Involvement in Pemphigus: A Literature Review. Biomed Res Int. 2018 Mar 25;2018:6154397. doi: 10.1155/2018/6154397. eCollection 2018. PMID 29770335
- [Background] Sar-Pomian M, Rudnicka L, Olszewska M. Trichoscopy - a useful tool in the preliminary differential diagnosis of autoimmune bullous diseases. Int J Dermatol. 2017 Oct;56(10):996-1002. doi: 10.1111/ijd.13725. Epub 2017 Aug 30. PMID 28856676
- [Background] Sar-Pomian M, Kurzeja M, Rudnicka L, Olszewska M. The value of trichoscopy in the differential diagnosis of scalp lesions in pemphigus vulgaris and pemphigus foliaceus. An Bras Dermatol. 2014 Nov-Dec;89(6):1007-12. doi: 10.1590/abd1806-4841.20143830. PMID 25387515
- [Background] Salmanpour R, Shahkar H, Namazi MR, Rahman-Shenas MR. Epidemiology of pemphigus in south-western Iran: a 10-year retrospective study (1991-2000). Int J Dermatol. 2006 Feb;45(2):103-5. doi: 10.1111/j.1365-4632.2004.02374.x. PMID 16445496
- [Background] Saleh MA, Ishii K, Yamagami J, Shirakata Y, Hashimoto K, Amagai M. Pathogenic anti-desmoglein 3 mAbs cloned from a paraneoplastic pemphigus patient by phage display. J Invest Dermatol. 2012 Apr;132(4):1141-8. doi: 10.1038/jid.2011.449. Epub 2012 Jan 26. PMID 22277944
- [Background] Rudnicka L, Olszewska M, Rakowska A, Slowinska M. Trichoscopy update 2011. J Dermatol Case Rep. 2011 Dec 12;5(4):82-8. doi: 10.3315/jdcr.2011.1083. PMID 22408709
- [Background] Rudnicka L, Olszewska M, Rakowska A, Kowalska-Oledzka E, Slowinska M. Trichoscopy: a new method for diagnosing hair loss. J Drugs Dermatol. 2008 Jul;7(7):651-4. PMID 18664157
- [Background] Rosenbach M, Murrell DF, Bystryn JC, Dulay S, Dick S, Fakharzadeh S, Hall R, Korman NJ, Lin J, Okawa J, Pandya AG, Payne AS, Rose M, Rubenstein D, Woodley D, Vittorio C, Werth BB, Williams EA, Taylor L, Troxel AB, Werth VP. Reliability and convergent validity of two outcome instruments for pemphigus. J Invest Dermatol. 2009 Oct;129(10):2404-10. doi: 10.1038/jid.2009.72. Epub 2009 Apr 9. PMID 19357707
- [Background] Rahbar Z, Daneshpazhooh M, Mirshams-Shahshahani M, Esmaili N, Heidari K, Aghazadeh N, Hejazi P, Ghajarzadeh M, Chams-Davatchi C. Pemphigus disease activity measurements: pemphigus disease area index, autoimmune bullous skin disorder intensity score, and pemphigus vulgaris activity score. JAMA Dermatol. 2014 Mar;150(3):266-72. doi: 10.1001/jamadermatol.2013.8175. PMID 24429657
- [Background] Pisanti S, Sharav Y, Kaufman E, Posner LN. Pemphigus vulgaris: incidence in Jews of different ethnic groups, according to age, sex, and initial lesion. Oral Surg Oral Med Oral Pathol. 1974 Sep;38(3):382-7. doi: 10.1016/0030-4220(74)90365-x. No abstract available. PMID 4528670
- [Background] Pirmez R. Acantholytic hair casts: a dermoscopic sign of pemphigus vulgaris of the scalp. Int J Trichology. 2012 Jul;4(3):172-3. doi: 10.4103/0974-7753.100087. PMID 23180929
- [Background] Murrell DF, Dick S, Ahmed AR, Amagai M, Barnadas MA, Borradori L, Bystryn JC, Cianchini G, Diaz L, Fivenson D, Hall R, Harman KE, Hashimoto T, Hertl M, Hunzelmann N, Iranzo P, Joly P, Jonkman MF, Kitajima Y, Korman NJ, Martin LK, Mimouni D, Pandya AG, Payne AS, Rubenstein D, Shimizu H, Sinha AA, Sirois D, Zillikens D, Werth VP. Consensus statement on definitions of disease, end points, and therapeutic response for pemphigus. J Am Acad Dermatol. 2008 Jun;58(6):1043-6. doi: 10.1016/j.jaad.2008.01.012. Epub 2008 Mar 14. PMID 18339444
- [Background] Kasperkiewicz M, Ellebrecht CT, Takahashi H, Yamagami J, Zillikens D, Payne AS, Amagai M. Pemphigus. Nat Rev Dis Primers. 2017 May 11;3:17026. doi: 10.1038/nrdp.2017.26. PMID 28492232
- [Background] Hennerici T, Pollmann R, Schmidt T, Seipelt M, Tackenberg B, Mobs C, Ghoreschi K, Hertl M, Eming R. Increased Frequency of T Follicular Helper Cells and Elevated Interleukin-27 Plasma Levels in Patients with Pemphigus. PLoS One. 2016 Feb 12;11(2):e0148919. doi: 10.1371/journal.pone.0148919. eCollection 2016. PMID 26872212
- [Background] Hebert V, Boulard C, Houivet E, Duvert Lehembre S, Borradori L, Della Torre R, Feliciani C, Fania L, Zambruno G, Camaioni DB, Didona B, Marinovic B, Schmidt E, Schumacher N, Hunefeld C, Schanz S, Kern JS, Hofmann S, Bouyeure AC, Picard-Dahan C, Prost-Squarcioni C, Caux F, Alexandre M, Ingen-Housz-Oro S, Bagot M, Tancrede-Bohin E, Bouaziz JD, Franck N, Vabres P, Labeille B, Richard MA, Delaporte E, Dupuy A, D'Incan M, Quereux G, Skowro F, Paul C, Livideanu CB, Beylot-Barry M, Doutre MS, Avenel-Audran M, Bedane C, Bernard P, Machet L, Maillard H, Jullien D, Debarbieux S, Sassolas B, Misery L, Abasq C, Dereure O, Lagoutte P, Ferranti V, Werth VP, Murrell DF, Hertl M, Benichou J, Joly P; French Study Group on Autoimmune Bullous Skin Diseases; Autoimmune Bullous Skin Disease Task Force of the European Academy of Dermatology and Venereology. Large International Validation of ABSIS and PDAI Pemphigus Severity Scores. J Invest Dermatol. 2019 Jan;139(1):31-37. doi: 10.1016/j.jid.2018.04.042. Epub 2018 Oct 6. PMID 30301637
- [Background] Hammers CM, Stanley JR. Mechanisms of Disease: Pemphigus and Bullous Pemphigoid. Annu Rev Pathol. 2016 May 23;11:175-97. doi: 10.1146/annurev-pathol-012615-044313. Epub 2016 Feb 22. PMID 26907530
- [Background] Fang H, Li Q, Wang G. The role of T cells in pemphigus vulgaris and bullous pemphigoid. Autoimmun Rev. 2020 Nov;19(11):102661. doi: 10.1016/j.autrev.2020.102661. Epub 2020 Sep 14. PMID 32942041
- [Background] Esmaili N, Chams-Davatchi C, Valikhani M, Daneshpazhooh M, Balighi K, Hallaji Z, Barzegari M, Akhyani M, Ghodsi ZS, Mrotazavi H, Naraghi ZS, Toosi S. Pemphigus vulgaris in Iran: a clinical study of 140 cases. Int J Dermatol. 2007 Nov;46(11):1166-70. doi: 10.1111/j.1365-4632.2007.03334.x. PMID 17988336
- [Background] David M, Katzenelson V, Hazaz B, Ben-Chetrit A, Sandbank M. Determination of IgG subclasses in patients with pemphigus with active disease and in remission. Arch Dermatol. 1989 Jun;125(6):787-90. PMID 2658844
- [Background] Daneshpazhooh M, Naraghi ZS, Ramezani A, Ghanadan A, Esmaili N, Chams-Davatchi C. Direct immunofluorescence of plucked hair for evaluation of immunologic remission in pemphigus vulgaris. J Am Acad Dermatol. 2011 Dec;65(6):e173-7. doi: 10.1016/j.jaad.2010.09.721. Epub 2011 Jun 22. PMID 21696851
- [Background] Berrih-Aknin S, Le Panse R. Myasthenia gravis: a comprehensive review of immune dysregulation and etiological mechanisms. J Autoimmun. 2014 Aug;52:90-100. doi: 10.1016/j.jaut.2013.12.011. Epub 2014 Jan 3. PMID 24389034
- [Background] Asothai R, Anand V, Das D, Antil PS, Khandpur S, Sharma VK, Sharma A. Distinctive Treg associated CCR4-CCL22 expression profile with altered frequency of Th17/Treg cell in the immunopathogenesis of Pemphigus Vulgaris. Immunobiology. 2015 Oct;220(10):1129-35. doi: 10.1016/j.imbio.2015.06.008. Epub 2015 Jun 17. PMID 26093920
- [Background] Arya SR, Valand AG, Krishna K. A clinico-pathological study of 70 cases of pemphigus. Indian J Dermatol Venereol Leprol. 1999 Jul-Aug;65(4):168-71. PMID 20921646
- [Background] Araghi F, Dadkhahfar S, Robati RM, Tabary M, Shahidi-Dadras M. The emerging role of T cells in pemphigus vulgaris: a systematic review. Clin Exp Med. 2023 Aug;23(4):1045-1054. doi: 10.1007/s10238-022-00855-8. Epub 2022 Aug 4. PMID 35925475